CLINICAL TRIAL: NCT06753617
Title: Safety and Feasibility of the Use of Cryoablation in Patients With Brain Tumors
Brief Title: Cryoablation of Brain Neoplasm
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Arnaud J.P.E. VIncent, Prof.dr, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NL81429.078.22
Record Dates: First submitted 2024-11-15; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Brain Neoplasm; Brain Metastases; Glioma; Meningioma
Keywords: Cryoablation; Cryosurgery; Brain neoplasm; Feasibility studies
MeSH Terms: conditions — Brain Neoplasms; Glioma; Meningioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cryoablation Treatment Group (Experimental): All patients enrolled in this study will undergo cryoablation as part of their surgical tumor resection procedure. The intervention will be integrated into the standard surgical approach.
  Interventions: Procedure: Cryoablation of brain neoplasm

INTERVENTIONS:
Procedure: Cryoablation of brain neoplasm — The procedure begins with standard surgical exposure of the tumor, followed by a biopsy. Next, one or more cryoprobes will be positioned directly into the tumor for ablation. Once positioned, the cryoablation process will commence. A maximum of 2x10 minutes cryoablation cycles will be established followed by active thawing. Following ablation, resection of the tumor will be performed, after which patients will receive standard treatment and follow-up care. Ice formation around the cryoprobes will be monitored using intraoperative ultrasound to optimize the ablation process.

SUMMARY:
This study will investigate the use of safety and feasibility of cryoablation in brain tumors

DETAILED DESCRIPTION:
Cryoablation is a therapeutic modality that employs extreme cold to induce cell necrosis in tumor tissue. While the application of cryoablation for the treatment of brain tumors remains under investigation, it has been extensively utilized in other organ systems with outcomes often surpassing those of conventional therapies.

The primary objective of this research is to evaluate the safety and feasibility of cryoablation as a treatment option for patients diagnosed with various brain tumors, including gliomas, meningiomas, and metastatic lesions. Participants enrolled in this study will first undergo standard surgical resection of the brain tumor. Prior to resection, a biopsy of the tumor will be performed to obtain a histopathological diagnosis, ensuring accurate characterization of the tumor type.

Subsequently, the tumor will undergo cryoablation utilizing cryoprobes, with a maximum of two cycles of up to 10 minutes each. The specific number and diameter of cryoprobes used will be determined by the tumor's size, aiming to achieve optimal ablation coverage. Following the removal of the cryoprobes, the tumor will be resected, and standard craniotomy closure procedures will be implemented. Patients will receive standardized postoperative care tailored to their clinical needs.

The follow-up period for this study will extend up to three months following the completion of treatment for the last enrolled participant, allowing for comprehensive assessment of treatment outcomes and safety profiles.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Tumor suspected as glioma (1. Astrocytoma, IDH mutant 2. Oligodendroglioma, IDH-mutant and 1p/19q-codeleted 3. Glioblastoma, IDH-wildtype), meningioma (WHO gr. 1 and gr 2), or brain metastasis based on preliminary diagnosis for which the patient will undergo surgery
* Supratentorial or infratentorial localization
* Safe trajectory/trajectories possible for ablation of at least 70% of the tumor, avoiding eloquent structures
* Karnofsky performance scale 70 or more
* Sufficient knowledge of the Dutch language to understand the study documents (in the judgement of the attending physician or researcher)
* Written Informed consent

Exclusion Criteria:

* <18 years or >80 years
* Tumor diameter bigger than 10 cm
* Unsafe trajectory (eloquent structures could be damaged)
* Pregnancy
* Contra-indication for general anesthesia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Safety: Incidence and Severity of Complications and Morbidity During the Study Period | From enrollment to the end of the study, with a minimum follow-up of 3 months. Complications such as bleeding, infection, epilepsy, brain edema, neurological deficit, and death will be evaluated, with safety assessed up to 12 months post-surgery.
  Complications & morbidity during the entire study period as decided by the treating physician. Severity and frequency of the following complications:
  * Postoperative intracranial bleeding
  * Wound infection
  * Epilepsy
  * Brain edema
  * Neurological deficit (paresis/plegia)
  * Aphasia
  * Death
Feasibility Evaluation in Operation Time | From start to end of the procedure, measured in minutes.
  Descriptive:
  Operation time (in minutes)
Feasibility Evaluation in Blood Loss | From start to end of the cryoablation procedure, measured in milliliters.
  Descriptive:
  Blood loss during intervention (in milliliters)

SECONDARY OUTCOMES:
Assessment of Tumor Cell Ablation: percentage of patients with total resections | For progression-free survival and overall survival, the time frame is defined as the period from the date of enrollment to 3 months after enrollment, with a minimum follow-up of 3 months.
  The percentage of patients with total resections (percentage of patients who undergo a complete tumor resection).
Assessment of Progression-Free Survival | From enrollment to 3 months after enrollment, with a minimum follow-up of 3 months.
  Progression-free survival (PFS) per patient, measured from the date of enrollment to 3 months after enrollment, assessed for disease progression or death.
Assessment of Overall Survival | From enrollment to 3 months after enrollment, with a minimum follow-up of 3 months.
  Overall Survival (OS) per patient type at 3 months, measured from the date of enrollment to 3 months after enrollment, assessed for survival (alive or deceased)

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Vincent, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-05): https://cdn.clinicaltrials.gov/large-docs/17/NCT06753617/Prot_SAP_000.pdf
  • Informed Consent Form (2024-01-05): https://cdn.clinicaltrials.gov/large-docs/17/NCT06753617/ICF_001.pdf